CLINICAL TRIAL: NCT06774209
Title: Multimodal PET Imaging in the Diagnosis and Treatment of Pelvic Tumors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PUMCH-NM-Pelvic Tumors-FAPI
Record Dates: First submitted 2024-10-17; First posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2024-10

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- imaging examinations (Experimental): The study recruited patients suffering from endometrial cancer, and three types of examinations will be performed on them.
  Interventions: Diagnostic Test: three kinds of examinations

INTERVENTIONS:
Diagnostic Test: three kinds of examinations — Following the enrollment of patients, both Gallium-68 labeled Fibroblast Activation Protein Inhibitor-04 Positron Emission Tomography/Computed Tomography (68Ga-FAPI-04 PET/CT) and Positron Emission Tomography/Magnetic Resonance Imaging (PET/MRI) scans are carried out. Additionally, within a one-week interval before and after the aforementioned examinations, Fluorine-18 labeled Fluorodeoxyglucose Positron Emission Tomography/Computed Tomography (18F-FDG PET/CT) is performed on the same cohort of patients.

SUMMARY:
This study is a prospective exploratory study to explore the application value of gallium 68 labeled-fibroblast activation protein inhibitor-04 Positron Emission Tomography（68Ga-FAPI-04 PET）imaging in patients with endometrial cancer and compare it with the imaging agent with better imaging effects to study its advantages. After patient enrollment, 68Ga-FAPI-04 Positron Emission Tomography/Computed Tomography（PET/CT） and Positron Emission Tomography/Magnetic Resonance Imaging（PET/MRI） examinations are performed, with the imaging agent administered intravenously at a dose of 0.02 to 0.04 mCi/Kg×patient weight (Kg), and a whole-body scan is performed 30-60 minutes later, with images processed as usual. Within 1 week before and after the examination, Fluorine18 labeled-Fluorodeoxyglucose Positron Emission Tomography/Computed Tomography（18F-FDG PET/CT） is completed, along with medical history collection and necessary laboratory tests. Subsequently, patients undergo surgical resection of the lesion and suspicious metastatic lymph nodes shown by FAPI PET/CT to obtain the corresponding pathological results. Finally, the diagnostic value of all patients in 68Ga-FAPI-04 PET/CT and PET/MR is analyzed and compared with 18F-FDG PET/CT to study the differences in diagnostic efficacy between the two.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years old
* Obtaining written informed consent
* Being able to accept follow-up
* Feasible surgery or biopsy to obtain the final result

Exclusion Criteria:

* Pregnant and lactating female patients
* Patients who are difficult to receive further diagnosis and treatment due to their severe condition
* Any patients with contraindications to magnetic resonance imaging

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
tumor size and SUVmax | Through study completion, an average of 1 year
  tumor size：unit（ Centimeter) Primary Tumor FAPI Uptake (SUVmax): This measures how much FAPI the primary endometrial cancer tumor takes up, using FAPI PET scans. It tells us how active the tumor cells are by comparing how much radiation the tumor tissue takes up compared to the normal tissue around it.

SECONDARY OUTCOMES:
Lymph Node Metastasis FAPI Uptake (SUVmax) and Distant Metastasis FAPI Uptake (SUVmax) | Through study completion, an average of 1 year
  Lymph Node Metastasis FAPI Uptake (SUVmax): This measures how much FAPI the lymph nodes that might have cancer spread to are taking up, using FAPI PET/CT scans. This helps us understand how active the cancer in the lymph nodes is.
  Distant Metastasis FAPI Uptake (SUVmax): This checks how much FAPI other cancer spots far from the lymph nodes are taking up. It helps us figure out how far the cancer has spread and how aggressive it is.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China